CLINICAL TRIAL: NCT02663414
Title: European Post-Market, Prospective, Multi-Center, Single-Arm Study to Evaluate Symptom Relief in Subjects With Medial Knee Osteoarthritis Treated With the Atlas Knee System for Load Reduction
Brief Title: European Post-Market Study for Medial Knee Osteoarthritis Treated With the Atlas Knee System for Load Reduction
Acronym: Atlas-PMCF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started and will never be started
Sponsor: Moximed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-102359
Record Dates: First submitted 2016-01-14; First posted 2016-01-26 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis (OA) of the Medial Knee Compartment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atlas device (Experimental): Each patient in this arm will receive the Atlas Knee System device on the medial side of the symptomatic knee.
  Interventions: Device: Atlas Knee System

INTERVENTIONS:
Device: Atlas Knee System — The Atlas Knee System is an approved device (CE Marked) and is an extra-capsular knee implant specifically designed to treat patients with uni-compartmental, medial knee osteoarthritis (OA).
  Other Names: Atlas System

SUMMARY:
The objective of this study is to collect post market data on safety and performance of the Atlas Knee System in patients with osteoarthritis (OA) of the medial knee compartment through a 24 months post-operative follow-up period.

DETAILED DESCRIPTION:
The objective of this study is to collect post market data on safety and performance of the Atlas Knee System in patients with osteoarthritis (OA) of the medial knee compartment through a 24 months post-operative follow-up period. This study is designed as a post-market, prospective, multicenter, single arm study. The study population will consist of adult subjects older than 25 years of age, with a diagnosis of symptomatic and radiographic OA of the medial knee compartment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, older than 25 years of age;
2. Have clinical symptoms in the study knee such as pain primarily localized to the medial aspect of the knee and generally exacerbated by weight bearing;
3. Radiographic confirmation of osteoarthritis of the medial knee compartment without bony erosion and best assessed using a Rosenberg view X-ray;
4. Have failed at least 6 months of conservative therapy prior to surgery with continued OA pain. Prior conservative therapy is defined as treatment including at least one of the following (OARSI Recommendations)9:

   1. Lifestyle modification;
   2. Weight loss, if BMI >35;
   3. Pain relievers;
   4. Physical therapy;
   5. Assist devices (Canes, Orthotics, Braces, etc.);
   6. Intra-articular (IA) injections.
5. Have active knee flexion ≥ 90⁰;
6. Are able to give voluntary, written informed consent to participate in this clinical investigation.
7. Are, in the opinion of the Clinical Investigator, able to understand this clinical investigation, cooperate with the investigational procedures, and are willing to return for all required post-treatment follow up visits.

Exclusion Criteria:

1. Clinical symptoms and radiographic evidence of OA in the lateral compartment of the study knee;
2. Clinical symptoms and radiographic evidence of OA in the patella-femoral compartment of the study knee;
3. Tibio-femoral alignment of > 10⁰ of varus, or > 6° of valgus, as measured using anatomical axis on a long standing (Hip-Knee-Ankle) antero-posterior (AP) view X-ray, or tibio-femoral alignment of > 16⁰ of varus, or > 0⁰ of valgus as measured using mechanical axis on a long standing (Hip-Knee-Ankle) AP view X-ray;
4. Previous joint modifying surgery in the study knee within 12 months prior to planned surgery date such as ligament reconstruction, meniscus repair, cartilage transplantation, and microfracture;
5. Arthroscopic surgeries for joint lavage, medial meniscectomy, chondral debridement, and loose body removal if within 3 months prior to planned surgery date; Note: concomitant diagnostic arthroscopy including debridement during Atlas procedure is permitted.
6. Active infection, sepsis, osteomyelitis or history of septic arthritis in any joint;
7. Rheumatoid arthritis, other forms of inflammatory joint disease or autoimmune disorder;
8. Excessive scarring of soft tissue structures of the medial knee;
9. Hyperextension > 10⁰;
10. Pathologic ligamentous instability (> 1 Medial collateral ligament injury or Lachman > 1 without hard stop) as assessed by the Investigator on physical examination;
11. Severe deformities leading to impaired fixation or improper positioning of the implant;
12. Paget's disease or metabolic disorders which may affect bone formation;
13. Known or suspected diagnosis of Osteomalacia;
14. Known or suspected diagnosis of Osteonecrosis;
15. Known or suspected diagnosis of Osteoporosis;
16. Rapid joint destruction, marked bone loss or bone resorption apparent on X-ray;
17. Charcot's joint disease or other severe neurosensory deficits;
18. Vascular insufficiency, muscular atrophy, neuromuscular disease;
19. Immunologically suppressed or immunocompromised;
20. History of systemic steroid treatment, medication use that affects bone metabolism (such as chemotherapy) within the previous 6 months, or radiotherapy within the previous 6 months;
21. Any significant medical condition and other factors that the investigator feels would interfere with the participation and completion of the study;
22. Pregnancy;
23. Subjects who are currently enrolled in another clinical investigation that could affect the results of this investigation.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Pain | Baseline and 24 month
  Change from baseline to 24 months in pain measured by the Knee injury and Osteoarthritis outcome score (KOOS).
Function | Baseline and 24 month
  Change from baseline to 24 months in patients functional outcome using the Knee injury and Osteoarthritis outcome score (KOOS).
Knee range of motion | Baseline and 24 month
  No change from baseline to 24 months in Knee range of motion as measured by Investigator Orthopedic examination.
Monitoring of adverse events | Baseline to 24 month
  Type, frequency, severity, and relatedness of adverse events will be assessed throughout the study.

SECONDARY OUTCOMES:
Function | Baseline and 24 month
  Change from baseline to 24 months in patients functional outcome measured by the Knee Society score (KSS).
Activity | Baseline and 24 month
  Change from baseline to 24 months in patients activity level using the University of California, Los Angeles (UCLA) activity scale.
Health outcome | Baseline and 24 month
  Change from baseline to 24 months in patients health outcome using a health outcome measure (EQ-5D).

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Yamut, Study Chair — Moximed